CLINICAL TRIAL: NCT06721676
Title: A Prospective, Single-center, Single-group Follow-up Study of Transcatheter Aortic Valve Replacement With A² Flex and Commissural Alignment Technology in Severe Aortic Stenosis by Peijia Medical
Brief Title: Study of Transcatheter Aortic Valve Replacement With A² Flex and Commissural Alignment Technology in Severe Aortic Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-496
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Aortic Stenosis Symptomatic
Keywords: aortic stenosis; TAVI; TAVR; Function of bending
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Transcatheter aortic valve system 2.5 generation is a new self-expanding valve system developed by Peijia Medical. Through the improvement of the delivery device to achieve A2 flex and commissural alignment technology, it can better manage the whole life cycle of AS patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single arm study (Experimental): The experimental apparatus consisted of artificial aortic valve, transporter and grip-loading system.the transporter has A2 flex function to improve coaxiality and commissural aligment to reduce coronary occlusion
  Interventions: Device: transcatheter aortic valve replacement in severe aortic stenosis

INTERVENTIONS:
Device: transcatheter aortic valve replacement in severe aortic stenosis — transcatheter aortic valve replacement with A² Flex and commissural alignment technology in severe aortic stenosis

SUMMARY:
A prospective, single-center, single-group follow-up study of transcatheter aortic valve replacement with A² Flex and commissural alignment technology in severe aortic stenosis by Peijia Medical

DETAILED DESCRIPTION:
A prospective, single-center, single-group follow-up study of transcatheter aortic valve replacement with A² Flex and commissural alignment technology in severe aortic stenosis by Peijia Medica.Patients are seen at pre and post procedure, discharge, 30 days. The main follow-up included clinical symptoms and signs, cardiac ultrasound, CT, etc. The outcome include immediate device success, procedure success and device sucess. The secondary end points include ：1) Immediate postoperative ultrasound evaluation of different sinus valve implantation depths.2) realization rate of commissural alignment was evaluated by ultrasound immediately after operation.3) the incidence of ≥ moderate paravalvular regurgitation assessed by ultrasound at 30 days after surgery.

4) CT assessment of different sinus valve implantation depths at 30 days after surgery.5) CT was performed 30 days after operation to evaluate the realization rate of commissural alignment and coronary artery alignment

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to participate and sign the informed consent and can cooperate with the whole trial process;
* Age ≥60 years old;
* Patients with severe calcified aortic stenosis confirmed by echocardiography (trans-aortic valve flow velocity ≥ 4.0m /s, or trans-active valvular pressure difference ≥40mmHg (1mmHg=0.133kPa), or aortic valve orientation area < 0.8cm2, or effective aortic valve orifice the product index is < 0.5cm2/m2);
* The cardiac team (at least two specialists in cardiovascular surgery) assessed the patient as unsuitable for routine surgery ;
* The aortic angel ≥60 degree.

Exclusion Criteria:

* The left and right coronary ostiums originate from the junctional zone or from both coronary ostiums;
* previous CABG history;
* Coronary ostial lesions（PCI or not）;
* Prior aortic valve prosthesis implantation (interventional/surgical, bioprosthetic/mechanical);
* Spoor peripheral arterial condition precluded transfemoral TAVR;
* Severe coronary stenoses requiring intervention for which concomitant PCI is not possible;
* Concomitant diseases requiring cardiac surgery;
* Other serious diseases that may reduce life expectancy to less than 12 months (e.g. clinically recurrent or metastatic cancer, congestive heart failure, etc.);
* contraindications to conventional cardiac catheterization, such as intracardiac thrombosis, infection, outflow obstruction, hypertrophic cardiomyopathy, etc;
* other surgical anatomical contraindications, such as the risk of coronary artery occlusion;
* clinically significant active bleeding
* platelet count < 30×10/ L;
* participating in other drug or medical device clinical studies that have not yet been completed ;
* considered inappropriate by the investigator to participate in the clinical study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Device success rate | at 30 days
  Device success is defined as - Vascular access, artificial aortic valve delivery and release were successful, and the delivery catheter was successfully withdrawn. - The artificial aortic valve was implanted in an anatomically accurate position. - The artificial aortic valve met the expected requirements (mean transvalvular pressure difference < 20mmHg or maximum flow rate < 3m/s; Doppler velocity index >_0.25,and less than moderate aortic regurgitation)

CONTACTS AND LOCATIONS:
Locations (1):
- Peiga Medical Technology (Suzhou) Co., Ltd, Suzhou, Jiangsu 215025, Suzhou, Jiangsu, China

REFERENCES:
- [Result] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Result] Vinayak M, Tang GHL, Li K, Berdan M, Koshy AN, Khera S, Lerakis S, Dangas GD, Sharma SK, Kini AS, Krishnamoorthy P. Commissural vs Coronary Alignment to Avoid Coronary Overlap With THV-Commissure in TAVR: A CT-Simulation Study. JACC Cardiovasc Interv. 2024 Mar 25;17(6):715-726. doi: 10.1016/j.jcin.2024.01.073. Epub 2024 Mar 6. PMID 38456886
- [Result] Bieliauskas G, Wong I, Bajoras V, Wang X, Kofoed KF, De Backer O, Sondergaard L. Patient-Specific Implantation Technique to Obtain Neo-Commissural Alignment With Self-Expanding Transcatheter Aortic Valves. JACC Cardiovasc Interv. 2021 Oct 11;14(19):2097-2108. doi: 10.1016/j.jcin.2021.06.033. Epub 2021 Sep 15. PMID 34538602